CLINICAL TRIAL: NCT07088029
Title: "Assessment of Occlusal Veneer Restorations Performance in Posterior Teeth Under Various Simulated Loading Conditions." (A 3D Finite Element Analysis Study)
Brief Title: Assessment of Occlusal Veneer Restorations Performance in Posterior Teeth
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: FDASU-Rec ID042514
Record Dates: First submitted 2025-06-15; First posted 2025-07-28 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Restoration of Posterior Teeth; Occlusal Veneers on Posterior Teeth
Keywords: occlusal veneer; direct occlusal veneer; clinical validation study; split-mouth clinical trial

STUDY DESIGN:
Intervention Model Description: Split-mouth design, one side (right/left posterior tooth) will be restored with a direct occlusal veneer (occlusal veneer of direct composite resin) and the other side (right/left posterior tooth) will restored with an indirect occlusal veneer (occlusal veneer of lithium disilicate).
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Direct occlusal veneer ( Occlusal Veneer of Composite resin) (Experimental): Split-mouth design, (right/left posterior tooth) will be restored with an occlusal veneer composite resin (Direct occlusal veneer). Directly fabricated occlusal veneers are a conservative approach, however, it requires a great skill from the operator to assure good margins and occlusal anatomy. Direct veneers are fabricated from composite resin and can be finished in a single visit, but longer chair time is required, in addition to the low wear resistance compared to ceramics. However, direct occlusal veneers have the benefit of resiliency close to that of natural dental tissue.
  Interventions: Procedure: Direct occlusal veneer ( Occlusal Veneer of Composite resin)
- Indirect occlusal veneer (Occlusal veneer of lithium disilicate) (Active Comparator): Split-mouth design, (right/left posterior tooth) will be restored with an Indirect occlusal veneer (Occlusal veneer of lithium disilicate). Indirectly fabricated occlusal veneers of lithium disilicate allow better control and design of the occlusal anatomy and proximal contacts, in addition to possessing better mechanical properties and fracture strength when compared to direct occlusal veneers. However, indirect occlusal veneers are lab fabricated, consequently, more clinical visits are required.
  Interventions: Procedure: Indirect occlusal veneer (Occlusal veneer of lithium disilicate)

INTERVENTIONS:
Procedure: Indirect occlusal veneer (Occlusal veneer of lithium disilicate) — Split-mouth design, (right/left posterior tooth) will be restored with an Indirect occlusal veneer (Occlusal veneer of lithium disilicate). Indirectly fabricated occlusal veneers of lithium disilicate allow better control and design of the occlusal anatomy and proximal contacts, in addition to possessing better mechanical properties and fracture strength when compared to direct occlusal veneers. However, indirect occlusal veneers are lab fabricated, consequently, more clinical visits are required.
  Other Names: Occlusal veneer of lithium disilicate
  Arms: Indirect occlusal veneer (Occlusal veneer of lithium disilicate)
Procedure: Direct occlusal veneer ( Occlusal Veneer of Composite resin) — Split-mouth design, (right/left posterior tooth) will be restored with an occlusal veneer composite resin (Direct occlusal veneer). Directly fabricated occlusal veneers are a conservative approach, however, it requires a great skill from the operator to assure good margins and occlusal anatomy. Direct veneers are fabricated from composite resin and can be finished in a single visit, but longer chair time is required, in addition to the low wear resistance compared to ceramics. However, direct occlusal veneers have the benefit of resiliency close to that of natural dental tissue.
  Other Names: Occlusal Veneer of Composite resin
  Arms: Direct occlusal veneer ( Occlusal Veneer of Composite resin)

SUMMARY:
The aim of the research is to study the mechanical behavior and clinical performance of veneers in posterior teeth. Clinical assessment and experimentation of two types of occlusal veneers will be conducted to evaluate their behavior.

DETAILED DESCRIPTION:
Occlusal veneers are restorations that restore the occlusal surface without axial wall involvement, allowing restoration of form, function, and esthetics of compromised or destroyed occlusal tooth structure in a conservative way as part of their treatment plan and the restorative process. The performance of occlusal veneer restorations is of paramount importance, as it determines the outcome and behavior of the final restoration. No ideal study has been conducted to evaluate teeth restored with occlusal veneer restorations. Evaluation must include all aspects of clinical performance, as some of the materials used in their fabrication have not been fully studied and should be studied to evaluate their clinical behavior using modified USPHS (United States Public Health Service) criteria. Which includes surface texture, anatomical form/wear, marginal integrity, marginal discoloration, secondary caries, color match and post-operative hypersensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Normal occlusion
* 25-35 years old
* Males or females having class II cavities indicated for occlusal veneers

Exclusion Criteria:

* Parafunctional habits
* Abnormal occlusion
* Extremely high caries risk patients
* Temporomandibular problems

Ages: 25 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Clinical assessment | 1 year follow up
  Clinical performance of each direct & indirect occlusal veneer using modified USPHS (United States Public Health Service) criteria. Each criterion will be graded as either Alpha, Bravo and Charlie.
  * Surface texture: aplha: smooth as surrounding enamel, beta: rougher than enamel, charlie: very rough
  * Anatomical wear; alpha: Restoration is continuous with existing tooth anatomy, bravo: Restoration is slightly discontinuous, charlie: restoration is discontinuous.
  * Marginal integrity: alpha: Closely adapted, beta: Visible crevice,, charlie Crevice in which dentin is exposed.
  * Marginal discoloration: alpha: No discoloration, bravo: Superficial staining , charlie: Deep staining.
  * Secondary caries: aplha: no caries, charlie: caries present.
  * Color match: aplha:No mismatch between restoration and tooth. bravo: Slight mismatch, charlie: unacceptable mismatch
  The clinical performance will be evaluated by blinded evaluators, the data will be collected in a table for analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Ain Shams University, Cairo, Heliopolis, Egypt

IPD SHARING:
Plan to Share IPD: No